CLINICAL TRIAL: NCT03179202
Title: A Post-Market Study of Percutaneous Peripheral Nerve Stimulation (PNS) for the Treatment of Back Pain
Brief Title: Electrical Stimulation for the Treatment of Back Pain Using Peripheral Nerve Stimulation (PNS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0142-CSP-000
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Back Pain; Low Back Pain
Keywords: Electrical Stimulation; Neurostimulation; Neuromodulation; Back Pain; Low Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Peripheral Nerve Stimulation (Experimental): All study subjects will have up to 4 Leads placed in their low back, will use the SPRINT Peripheral Nerve Stimulation (PNS) System, and will receive electrical stimulation.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT PNS System is a device which delivers mild electrical stimulation to the muscles in the low back. The System includes up to four small wires (called "Leads") that are placed through the skin into the muscles in the low back. The wires attach to device(s) worn on the body that deliver stimulation (called Stimulators). The PNS System was approved by the FDA for up to 60 days of use for the management of acute and chronic pain, including back pain.
  Other Names: SPRINT System; Smartpatch System; SPRINT; Smartpatch

SUMMARY:
The purpose of this study is to evaluate the effectiveness of electrical stimulation (low levels of electricity) on low back pain. This study involves the SPRINT Peripheral Nerve Stimulation (PNS) system. The System delivers mild electrical stimulation to the nerves in the low back. The System includes up to four small wires (called "Leads") that are placed through the skin into the muscles in the low back. The wires attach to device(s) worn on the body that deliver stimulation (called Stimulators).

ELIGIBILITY:
Key Inclusion Criteria:

* At least 21 years of age
* Chronic low back pain

Key Exclusion Criteria:

* Infection on or around the low back
* Conditions with increased risk of infection (e.g., valvular heart disease, compromised immune system, history of recurrent skin infections)
* Implanted electronic device
* Body Mass Index (BMI) > 40
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Hope Research Institute, Peoria, Arizona
  - Integrated Pain Management Medical Group, Walnut Creek, California
  - International Spine, Pain and Performance Center, Washington D.C., District of Columbia
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Virginia iSpine Physicians, Richmond, Virginia
  - The Spine and Nerve Center of St. Francis Hospital, Charleston, West Virginia

REFERENCES:
- [Derived] Gilmore CA, Deer TR, Desai MJ, Li S, DePalma MJ, Cohen SP, Swan BD, McGee MJ, Boggs JW. Four-Year Follow-Up from a Prospective, Multicenter Study of Percutaneous 60-Day Peripheral Nerve Stimulation for Chronic Low Back Pain. Pain Ther. 2025 Jun;14(3):1103-1115. doi: 10.1007/s40122-025-00737-3. Epub 2025 Apr 22. PMID 40261580
- [Derived] Deer TR, Gilmore CA, Desai MJ, Li SC, DePalma MJ, Hopkins TJ, Burgher AH, Spinner DA, Cohen SP, McGee MJ, Boggs JW. Percutaneous Peripheral Nerve Stimulation of the Medial Branch Nerves for the Treatment of Chronic Axial Back Pain in Patients After Radiofrequency Ablation. Pain Med. 2021 Mar 18;22(3):548-560. doi: 10.1093/pm/pnaa432. PMID 33616178
- See also: Sponsor's Website — http://www.sprtherapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in June 2017 and was concluded in December 2019. Subjects were screened from the available pool of candidates who presented with chronic low back pain.
Pre-assignment Details: After obtaining informed consent, subjects were evaluated for eligibility.
Groups:
- Consented Subjects: Subjects who signed an informed consent form.
Period: Overall Study
Arm/Group | Consented Subjects
Started | 166
Enrolled/Received Leads (Subjects who were consented, met eligibility criteria, and underwent Lead Placement. Also includes subjects participating in sub-studies with modified eligibility criteria allowing a history of prior radiofrequency ablation or prior lumbar surgery.) | 99
Protocol Population (Subjects who were consented, met eligibility criteria, underwent Lead Placement, and continued to meet eligibility criteria. Also includes subjects participating in sub-studies with modified eligibility criteria allowing a history of prior radiofrequency ablation or prior lumbar surgery.) | 91
Completed | 75
Not Completed | 91
Not completed — Screen Failure | 67
Not completed — Subject Lost to Follow Up | 12
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 3
Not completed — Unrelated Death Reported in All-Cause Mortality | 1
Not completed — Other Reason: Incarceration after Enrollment | 1

BASELINE CHARACTERISTICS:
Groups:
- Enrolled/Received Leads: Subjects who were consented, met eligibility criteria, and underwent Lead placement. Also includes subjects participating in sub-studies with modified eligibility criteria allowing a history of prior radiofrequency ablation or prior lumbar surgery.
Arm/Group | Enrolled/Received Leads
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 84
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 99
Duration of Low Back Pain [Mean (Standard Deviation); unit: years] | 17.2 (14.7)
Employment Status [Count of Participants; unit: Participants]
  Currently Working | 44
  On Leave of Absence | 1
  Retired (not due to health) | 30
  Homemaker | 4
  Unemployed | 7
  Student | 2
  Disabled and/or Retired Because of Low Back Pain | 8
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Experienced ≥30% Reduction in Average Low Back Pain Intensity
Description: All subjects were asked to complete daily diaries to record their average pain intensity on each day of a 7-day period. The pain intensity question was excerpted from the Brief Pain Inventory-Short Form Question 5 (BPI-5). The BPI-5 uses an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." For each subject, the mean score for the baseline and end of treatment (EOT) diary periods were calculated and percent reduction was determined. Subjects that achieved ≥30% reduction in pain, were considered successful.
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. EOT data were not available for eight subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Protocol Population: Subjects who were consented, met eligibility criteria, underwent Lead Placement, and continued to meet eligibility criteria. Also includes subjects participating in sub-studies with modified eligibility criteria allowing a history of prior radiofrequency ablation or prior lumbar surgery.
Arm/Group | Protocol Population
Number analyzed (Participants) | 83
Participants | 58

2. Primary Outcome: Number of Subjects That Experienced at Least One Study-Related Adverse Event
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition has occurred since their previous visit. If the subject experienced a change that was an adverse event, an Adverse Event Form was completed by the site. The number of subjects that experienced at least one study-related adverse event is reported here.
Time Frame: Up to 15 months for each subject from baseline to the last study visit
Population: All enrolled subjects that received leads are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled/Received Leads
Number analyzed (Participants) | 99
Participants | 49

3. Secondary Outcome: Worst Pain Intensity
Description: All subjects were asked to complete daily diaries to record their worst pain intensity on each day of a 7-day period. The pain intensity question was excerpted from the Brief Pain Inventory-Short Form Question 3 (BPI-3). The BPI-3 uses an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." For each subject, the mean score for the baseline and end of treatment (EOT) diary periods were calculated. The mean score across all subjects for each time point is reported.
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. EOT data were not available for eight subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol Population
Number analyzed (Participants) | 91
score on a scale
  Baseline | 7.7 (1.2)
  EOT: number analyzed (Participants) | 83
  EOT | 4.5 (2.1)

4. Secondary Outcome: Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) is a widely used assessment designed to measure the degree of disability in people with low back pain. This validated questionnaire includes topics concerning the intensity of pain, the subject's ability to perform normal daily activities such as personal care, walking, sitting, or standing, and how pain affects the subject's sex life, social life, and travel. The scale ranges from 0-100 and higher scores indicate greater disability due to low back pain. The mean score across all subjects at baseline and end of treatment (EOT) is reported here.
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. Data were not available for one subject at baseline and for eight subjects at EOT.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol Population
Number analyzed (Participants) | 91
score on a scale
  Baseline | 39.1 (12.1)
  EOT: number analyzed (Participants) | 83
  EOT | 23.6 (12.6)

5. Secondary Outcome: Mean Change in Health-Related Quality of Life
Description: The RAND 36-Item Short Form Health Survey is a widely accepted form used to quantify quality of life. The survey consists of 8 categories with a total of 36 questions regarding the subject's general health and activities. The survey assesses physical and emotional problems associated with pain during the past 4 weeks. Each category is scored on a 0-100 scale, where a higher score indicates a more favorable health state. The score for each category was calculated at baseline and End of Treatment (EOT) for each subject. The change in each category score from Baseline to EOT was then calculated for each subject (with a positive change indicating an increase in health-related quality of life). The mean and standard deviation of the subjects' changes in each category are presented below.
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. Data were not available for three subjects at baseline and five subjects at end of treatment (EOT).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol Population
Number analyzed (Participants) | 88
score on a scale
  Physical Functioning | 13.2 (19.6)
  Role Limitations due to Physical Health | 26.6 (39.9)
  Role Limitations due to Emotional Problems | 12.2 (42.5)
  Energy/Fatigue | 12.8 (17.0)
  Emotional well-being | 7.2 (15.2)
  Social Functioning | 18.0 (22.5)
  Pain | 21.6 (20.8)
  General Health | 5.0 (15.1)

6. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory (BDI-II) is a validated, 21-question survey used to measure depression severity. Questions are rated on a scale from 0 to 3, and the scores from each question are totaled to provide an overall score ranging between 0 to 63. Scores from 0-13 indicate minimal depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 indicates severe depression. The average total scores across subjects were calculated at baseline and end of treatment (EOT).
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. EOT data were not available for nine subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol Population
Number analyzed (Participants) | 91
score on a scale
  Baseline | 8.9 (5.6)
  EOT: number analyzed (Participants) | 82
  EOT | 5.2 (5.1)

7. Secondary Outcome: Patient Global Impression of Change (PGIC) Survey
Description: The Patient Global Impression of Change (PGIC) asks subjects to rate their improvement with treatment on a 7-point scale where 1 represents "very much worse" and 7 represents "very much improved" as compared to before stimulation treatment. The subjects combine all the components of their experience into one overall score. The number of participants with each rating after 8 weeks of treatment is reported here.
Time Frame: 8-weeks post-Start of Treatment (SOT)
Population: Protocol Population presented. EOT data were not available for eight subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol Population
Number analyzed (Participants) | 83
Participants
  Very Much Improved | 12
  Much Improved | 39
  Minimally Improved | 23
  No Change | 8
  Minimally Worse | 0
  Much Worse | 1
  Very Much Worse | 0

8. Secondary Outcome: Pain Interference
Description: Question 9 of the Brief Pain Inventory-Short Form (BPI-9) is a 7-part question that assesses the level of interference that subjects experience in their daily lives due to pain. The 7 categories are general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Subjects were asked to rate how much their low back pain interferes with each aspect on an 11-point numerical scale where 0 represents "Does Not Interfere" and 10 represents "Completely Interferes." The average of these 7 scores was calculated for each subject. The mean was taken across subjects for each time point.
Time Frame: Baseline and End of Treatment (EOT= 8-weeks post-start of treatment)
Population: Protocol Population presented. Data were not available for nine subjects at end of treatment (EOT).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protocol Population
Number analyzed (Participants) | 91
score on a scale
  Baseline | 5.7 (2.0)
  EOT: number analyzed (Participants) | 82
  EOT | 2.8 (2.0)

ADVERSE EVENTS:
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through the 12-month follow up visit. The total assessment period was approximately 14 months for each participant.
Arm/Group | Enrolled/Received Leads
All-Cause Mortality (participants affected / at risk) | 1/99
Serious Adverse Events (participants affected / at risk) | 4/99
Other Adverse Events (participants affected / at risk) | 49/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled/Received Leads (N=99)
Shoulder procedure (Surgical and medical procedures) | 1 (1) — Not Study-Related
Heart attack (Cardiac disorders) | 1 (1) — Not Study-Related
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Study-Related
Heart procedures (Surgical and medical procedures) | 1 (2) — Not Study-Related
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Study-Related
Liver/Lymph node metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not Study-Related
SCS trial and permanent implant (Surgical and medical procedures) | 1 (1) — Not Study-Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled/Received Leads (N=99)
Irritation at pad and/or Lead exit sites (Skin and subcutaneous tissue disorders) | 16 (17) — Study-Related
Irritation or bruising at bandage site or connector cradles (Skin and subcutaneous tissue disorders) | 19 (19) — Study-Related
Mild swelling following Lead removal (Skin and subcutaneous tissue disorders) | 1 (1) — Study-Related
Generalized itching (Skin and subcutaneous tissue disorders) | 1 (1) — Unable to determine relationship to study
Itching at pad and/or Lead exit sites (Skin and subcutaneous tissue disorders) | 11 (11) — Study-Related
Itching at bandage site (Skin and subcutaneous tissue disorders) | 13 (13) — Study-Related
Discoloration/bruising at Lead exit site (Skin and subcutaneous tissue disorders) | 1 (1) — Study-Related
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2) — Study-Related
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — Study-Related
Discharge or bleeding from electrode/insertion site (Skin and subcutaneous tissue disorders) | 3 (3) — Study-Related
Granuloma (Skin and subcutaneous tissue disorders) | 2 (2) — Study-Related
Miscellaneous (Skin and subcutaneous tissue disorders) | 2 (2) — Study-Related
New leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Study-Related
Pain from Lead Placement (Musculoskeletal and connective tissue disorders) | 3 (3) — Study-Related
Pain/discomfort at lead site (Musculoskeletal and connective tissue disorders) | 5 (5) — Study-Related
Pain from stimulation (Musculoskeletal and connective tissue disorders) | 2 (3) — Study-Related
Uncomfortable stimulation (Musculoskeletal and connective tissue disorders) | 8 (8) — Six events were study-related and two event relationships were unable to be determined.
Worsening low back pain (Musculoskeletal and connective tissue disorders) | 4 (4) — One event was study-related, and three events were not related to the study.
Exacerbation of low back pain from medial branch block (Musculoskeletal and connective tissue disorders) | 1 (1) — Study-Related
Shoulder and/or hip conditions (Musculoskeletal and connective tissue disorders) | 3 (4) — Not Study-Related
Thoracic pain/hematoma from fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Not Study-Related
Pain (distal or unrelated to device location) (Musculoskeletal and connective tissue disorders) | 6 (6) — Five events were not related to the study and one event relationship was unable to be determined.
Shortness of breath (Cardiac disorders) | 1 (1) — Not Study-Related
Vasovagal dizziness following lead placement (Cardiac disorders) | 2 (2) — One event was study-related, and the other relationship was unable to be determined
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Not Study-Related
Bacterial pneumonia (General disorders) | 1 (1) — Not Study-Related
Strep throat (General disorders) | 1 (1) — Not Study-Related
Sinus infection (General disorders) | 2 (2) — Not Study-Related
Sinuplasty (Surgical and medical procedures) | 1 (1) — Not Study-Related
Toenail removal (Surgical and medical procedures) | 1 (1) — Not Study-Related
Shoulder procedure (Surgical and medical procedures) | 1 (1) — Not Study-Related
Hip procedure (Surgical and medical procedures) | 1 (1) — Not Study-Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03179202/Prot_SAP_001.pdf